CLINICAL TRIAL: NCT02727049
Title: Motion Capture and Analysis of NYIT Athletes
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no college athlete availability
Sponsor: New York Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BHS1064
Record Dates: First submitted 2015-02-12; First posted 2016-04-04 (Estimated); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Athletic Injuries
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- injured athlete for OMM (Experimental): Participating athletes who sustain an injury will receive standard of care with the Intervention osteopathic manipulative medicine (OMM)
  Interventions: Other: Osteopathic manipulative medicine (OMM)
- injured athlete no OMM (No Intervention): Participating athletes who sustain an injury will receive standard of care withOUT osteopathic manipulative medicine (OMM)

INTERVENTIONS:
Other: Osteopathic manipulative medicine (OMM) — Osteopathic manipulative medicine includes all types of manual therapies to gently restore and/or optimize one's natural joint, muscle, and other soft tissue balance.
  Other Names: osteopathic manual therapy
  Arms: injured athlete for OMM

SUMMARY:
The purpose of this research is to:

1. determine the normal or existing dynamic biomechanics of college athletes and
2. test the effectiveness of osteopathic manipulative medicine in the treatment of athletic injuries.

Motion capture using Vicon systems allows researchers to quantify characteristics of a body such as the range of motion of the hip or shoulder during an athletic technique such as kicking or shooting a basketball into the basket. The quantified information has been used before to better understand human mobility and performance. Osteopathic manipulative medicine (OMM) is manual medicine applied to joints, muscles, and connective tissue with a goal of improved body functions. Research demonstrating effectiveness of OMM on the musculoskeletal and associated connective tissue systems health includes, among others, prospective clinical trials of OMM for treatment of neck pain, low back pain, and acute first- and second-degree ankle sprains.

DETAILED DESCRIPTION:
Volunteers for the study will be recruited through their Athletic director, coach, or physician by an announcement made verbally or via email. The motion capture will be performed under Matthew Cornelius, MS using the Vicon Bonita Motion Capture system in the Fine Arts Department of NYIT. Following the motion capture, body biomechanics will be analyzed to determine the range of motion of each joint in sagittal, frontal, and horizontal planes as well as the timing and sequence of the movements. The motion analysis will be compared to the Sports Physical exam, including the general, structural/neuromusculoskeletal, and central neurological (ImPACT) exams. The comparison will add validity to the physical exam. In addition, determining if the quantitative, 3-dimensional motion analysis can be correlated with information from the physical exam with regards to restrictions to motion may be useful for athletes to optimize their abilities in the future. If during the course of the athlete's training and competition season s/he sustains an injury, s/he will be evaluated by the NYIT athletics physician, who will randomly assign the injured athletes to either the 'standard of care without OMM' or 'standard of care with OMM' cohorts when medically appropriate. OMM will be performed by an NYITCOM physician specializing in family medicine and OMT or neuromusculoskeletal systems and OMM. "Return to play' time and post-intervention/post-control quantitative motion analysis of biomechanics during the athletes demonstration of the same athletic maneuvers as before the injury.

ELIGIBILITY:
Inclusion Criteria:

* athlete at new York Institute of Technology
* approval by NYIT Athletics Physical for participation in sports
* no current injury

Exclusion Criteria:

* illness preventing participation in sports
* any current injury
* younger than 18 years of age
* pregnancy
* allergy to spandex, nylon, or polyester

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-02; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
change in joint angles (degrees) | 1 year
  quantitative biomechanical testing will be performed before and after OMM or control

CONTACTS AND LOCATIONS:
Overall Officials: Jayme D Mancini, DO PhD, Principal Investigator — New York Institute of Technology
Locations (2):
- United States (2):
  - New York Institute of Technology College of Osteopathic Medicine Academic Health Care Center, Old Westbury, New York
  - New York Institute of Technology, Old Westbury, New York

IPD SHARING:
Plan to Share IPD: No